CLINICAL TRIAL: NCT02726854
Title: Apatinib as Second-line Treatment of Advanced Pancreatic Cancer, Phase II Clinical Study of Open Arm
Brief Title: Apatinib as Second-line Treatment of Advanced Pancreatic Cancer
Acronym: Apslpanc
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-024
Record Dates: First submitted 2016-03-16; First posted 2016-04-04 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib (Experimental): Patients will be offered with Apatinib (850mg daily,orally)until their disease have progressed.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Patients with pancreatic cancer who are failed of receiving first-line chemotherapy and cannot tolerate second-line chemotherapy or unwilling to receive second-line chemotherapy will receive Apatinib Tablets (850mg once daily, orally) 30 minutes after meal with warm water. Take 28 days as a cycle, patients will receive this treatment until they have got disease progressed.
  Other Names: YN968D1

SUMMARY:
The main research purpose Evaluation of objective response Apatinib second-line treatment of advanced pancreatic cancer (ORR) and the rate of progression free survival (PFS).

Objective to study the objective and exploratory secondary research To observe the Apatinib in second line treatment of advanced pancreatic cancer disease control rate (DCR), patients with overall survival (OS) benefit, treatment effects on quality of life (QOL) score and drug safety evaluation, To investigate the relationship of apatinib as second-line treatment of advanced pancreatic cancer and the expression of vascular endothelial growth factor receptor(VEGFR) in the serum

DETAILED DESCRIPTION:
The purpose of this study is to determine what effects apatinib has on advanced pancreatic cancer patients after failure of first-line chemotherapy cannot tolerate second-line chemotherapy or unwilling to receive second-line chemotherapy of pancreatic cancer patients.To investigate the relationship between apatinib as second-line treatment of advanced pancreatic cancer and the expression of vascular endothelial growth factor receptor(VEGFR) in the serum.

This study choose the First Affiliated Hospital of Xi'an JiaoTong University were unable to tolerate the failure of first-line chemotherapy for second-line chemotherapy or unwilling to receive second-line chemotherapy of pancreatic cancer patients as the research object, the clinical data of clinical subjects age and sex, Eastern Cooperative Oncology Group （ECOG） score, tumor stage, pathological type, pathological grading, giving apatinib treatment, during the treatment of blood monitoring in patients with CA199 levels, imaging findings, assessment of tumor related symptoms and adverse events, and the expression of VEGFR in blood was measured by ELISA method, the curative effect evaluation of the end of the 2 cycle of treatment, patients with effective evaluation to oral apatinib, through the statistical analysis of the data of complete remission (CR) or partial remission (PR), the rate of progression free survival (PFS) expression of CA199 content in serum and serum VEGFR levels of the relevant indicators,. Explore Apatinib for the curative effect and safety of the second-line treatment of advanced pancreatic cancer, and to explore the relationship between the serum VEGF expression level.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age,Male or female;
* The advanced pancreatic cancer pathology, with measurable lesions (spiral CT scan is more than 10mm, according to the standard of RECIST 1.1);
* Locally advanced, unresectable recurrent or metastatic pancreatic cancer;
* According to CTCAE 4.0 and patient complaints, the researchers determine second-line chemotherapy should not be tolerated by the patients or patients want to receive second-line chemotherapy.
* ECOG performance scale 0-1;
* Baseline blood routine and biochemical indexes meet the following criteria:
* Hemoglobin ≥ 80g/L,
* The absolute neutrophil count (ANC) ≥ 1.5 ×109/L,
* Blood platelet ≥ 90 ×109/L
* Alanine aminotransferase(ALT),Aspartate transaminase (AST) less than 2.5 times the upper limit of normal value, equal to or less than 5 times the upper limit of normal (liver metastasis),
* the serum total bilirubin is less than 1.5 times the upper limit of normal value,
* Serum creatinine. Less than 1.5 times the upper limit of normal value,
* Serum albumin is more than 30g/L;
* Life expectancy ≥ 3 months.
* women of childbearing age to within 7 days before entering the group of serum or urine pregnancy test and the results were negative. And be willing to give drug test during the test and the last 8 weeks using an appropriate method of contraception. For men, for sterilization, or agreed to during the period of the experiment and at the end of the given experimental drugs for 8 weeks by appropriate methods of contraception;
* In this study, volunteer subjects signed the informed consent, good compliance with follow-up.

Exclusion Criteria:

* It is confirmed that of apatinib and / or its accessories allergy;
* Have high blood pressure and antihypertensive drug treatment can not drop to normal range(systolic pressure >140 mmHg, diastolic blood pressure 90>mmHg), suffering from coronary artery disease above grade I, grade I arrhythmia (including corrected QT interval prolongation male > 450 ms, women > 470 MS) and grade I heart insufficiency; urine protein positive patients.
* Has a variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.);
* Coagulant function abnormality (INR>1.5, activated partial thromboplastin time(APTT)>1.5, ULN) with bleeding tendency;
* patients with central nervous system metastasis;
* pregnant or lactating women;
* Patients with other malignant tumors within five years;
* Has a history of psychiatric drugs abuse and can't quit or patients with mental disorders;
* 4 weeks participated in other clinical trials of patients;
* received VEGFR inhibitors, such as sorafenib, chougny for treatment;
* According to the researcher's judgment, there is serious to endanger the safety of patients or affect patients with disease to do the research;
* The researchers think that the person doesn't fit into.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
PFS(Progression free survival) | 8 Weeks
ORR (Objective response rate) | 8 Weeks

SECONDARY OUTCOMES:
DCR(disease control rate) | 8 Weeks
OS (Overall survival) | 8 Weeks
QoL (Quality of life as assessed by EORTC QLQ-C30） | 8 Weeks
Number of participants with treatment-related adverse events as assessed by NCI-CTC（V3.0） | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enxiao Li, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First affiliate hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided